CLINICAL TRIAL: NCT00490464
Title: Safety and Efficacy of Nicardipine for the Control of Blood Pressure After SAH
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Other Study IDs: 2004-0233
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Subarachnoid Hemorrhage; Intracerebral Hemorrhage
Keywords: Patients with SAH or ICH
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage; Hepatitis, Infectious Canine | interventions — Nicardipine; Nitroprusside

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nicardipine and Nipride

SUMMARY:
The purpose of this research is to explore ways to improve and simplify control of blood pressure in patients with SAH or ICH. This research will be done by comparing tow different medications that are routinely used to help control blood pressure. None of the medications used in this study nor any procedures performed are experimental.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old (inclusive)
* Admission to NSICU with a diagnosis of SAH or ICH

Exclusion Criteria:

* Patients who are admitted >48 hours after SAH or ICH
* Readmission or second SAH
* Readmission or second ICH
* Large (immediately life threatening) associated intraparenchymal or intraventricular hemorrhage
* Women who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2004-06; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Z Roitberg, MD, Principal Investigator — University of Illinois at Chicago, Department of Neurosurgery
Locations (1):
- University of Illinois at Chicago, UIC, Chicago, Illinois, United States